CLINICAL TRIAL: NCT03523455
Title: The Effects of Iron Aid IPS on Performance, Fatigue and Iron Levels During 12 Weeks of Supplementation and Aerobic Training
Brief Title: Iron Aid IPS on Performance, Fatigue and Iron Levels During 12 Weeks of Supplementation and Aerobic Training
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit qualified participants
Sponsor: University of Mary Hardin-Baylor (Other)
Collaborators: ChemiNutra (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRA-1
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Iron-deficiency
Keywords: Iron; Exercise Performance; Fatigue
MeSH Terms: conditions — Anemia, Iron-Deficiency; Fatigue | interventions — iron protein succinylate; Sugars

STUDY DESIGN:
Intervention Model Description: Two groups: placebo, 30mg dose
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Maltodextrin (matches the weight of the active treatment) Taken once each day after breakfast, but before lunch.
  Interventions: Other: Sugar Pill
- Iron Aid IPS (Iron Protein Succinylate) (Active Comparator): IronAid Iron Protein Succinylate 30 mg Taken once each day after breakfast, but before lunch.
  Interventions: Dietary Supplement: Iron Aid IPS (Iron Protein Succinylate)

INTERVENTIONS:
Dietary Supplement: Iron Aid IPS (Iron Protein Succinylate) — Taken orally in capsule form
  Arms: Iron Aid IPS (Iron Protein Succinylate)
Other: Sugar Pill — Taken orally in capsule form
  Arms: Sugar Pill

SUMMARY:
Participants are required to undergo a screening and qualification before beginning the study. Once qualified, baseline testing is completed in the laboratory. This testing includes: body composition measurements, a blood draw, questionnaires, a VO2 max test, and a time to exhaustion trial. This testing is repeated during week 4 and week 12. At week 8, subjects complete a blood draw and questionnaires only. During the 12 week period, participants will follow an endurance exercise program in which they will train 4 days per week. This is a double-blind study in which participants are randomized into either the placebo or supplement group. They are instructed to ingest the supplement once a day at breakfast. Diet logs are also monitored throughout the duration of the study with the restriction of no red meat.

DETAILED DESCRIPTION:
Subjects expressing interest in participating in this study, were interviewed in person to determine whether they appeared to qualify to participate in the study. If they met eligibility criteria, they were invited to attend an entry/familiarization session. During this session, they completed personal and medical histories which were reviewed to determine whether they met eligibility criteria. Once meeting entry criteria, they were familiarized to the study protocol via a verbal and written explanation outlining the study design. Subjects then read and signed the Informed Consent Statements after the study details were explained. Subjects then perform the exercise protocol in which they must have completed in order to qualify for the study.

Subjects were asked to perform a VO2 Max test using the Bruce protocol. Following the VO2 Max test, subjects were given a rest period of 20 minutes before starting the Time to Exhaustion (TTE) trial run. This session familiarized subjects with the exercise protocol preparing them for the qualification testing session. Subjects then returned to the lab in a 12 hour fasted state and completed a VO2max test. If a 42 ml/kg/min or above was achieved subjects were then allowed to complete the 20 minute TTE test. After completion of the TTE, a blood draw was done to access the subject's iron levels. Once results for iron levels returned at a 90 or below subjects were given an appointment time to perform baseline assessments and testing sessions.

Baseline testing (Week 0), Week 8 and Week 12 took place on the 8th or 9th day after the subject's menstrual cycle. Subjects returned to the lab in a 12 hour fasted state, with no strenuous workouts done 48 hours prior to testing. Subjects had their height and weight measured, filled out questionnaires, completed a DEXA scan and InBody to establish current body composition, afterwards having their heart rate and blood pressure assessed. At this point subjects were instructed to lay on a table for their blood draw. Once the blood draw was done, subjects completed a VO2 Max test using the Bruce protocol. Following the VO2 Max testing, subjects filled out 2 questionnaires and were given a rest period of 20 minutes before starting the Time to Exhaustion (TTE) trial run. During the rest period subjects were given a snack to ingest (banana or apple) and consumed the same snack at each testing session. Approximately 12 minutes prior to the TTE subjects filled out a questionnaire. During the TTE run subjects were able to control and see the speed at which they ran but were blinded to the time passed along with the distance completed. After the 20 minutes, the treadmill stopped, distance, heart rate and blood pressure were measured. Afterwards, subjects filled out post exercise questionnaires. At week 0, after all exercise testing was completed, subjects were assigned to a group (either placebo or active) and instructed to ingest 1 capsule per day. A workout log was also provided to each subject, who would return to the lab every Friday with their workout log to access exercise compliance.

At week 4, subjects returned to the lab on the 8th or 9th day after their menstrual cycle to have a blood draw completed to access blood marker variables in addition to questionnaires.

Diet logs were keep throughout the duration of the study and were monitored by lab staff.

ELIGIBILITY:
Inclusion Criteria:

1. I am willing to and provide written and dated informed consent form to participate in the study;
2. I am female 18-30 years of age;
3. I am willing and able to comply with protocol;
4. My VO2 max is in compliance with age range (42 ml/kg/min);
5. I have not used or consumed any prescription drugs or supplements that could potentially confound the results of the current supplement;
6. I am apparently healthy and free from disease, as determined by a health history questionnaire;
7. I agree to abstain from strenuous activity and pre-workout supplementation 48 hours prior to each testing visit;
8. I must be fasted for 8 hours prior to each testing visit;
9. I agree to abstain from caffeine and alcohol consumption 24 hours prior to each testing visit;
10. I do not have any existing muscular disorders;
11. I am able to complete all testing on the 8th or 9th day after my menstrual cycle has ended.

Exclusion Criteria:

1. I use tobacco products or have quit within the past 6 months;
2. I am currently pregnant, plan on becoming pregnant, or become pregnant during the duration of the study;
3. I have given birth or been pregnant the past year;
4. I am currently taking or have taken any oral contraception within the past 6 months;
5. I have difficulty giving blood;
6. I am currently diagnosed with having or currently involved in a managed treatment plan for any known metabolic disorder including heart disease, arrhythmias, diabetes, gall bladder, thyroid disease, or hypogonadism;
7. I am diagnosed with having or are currently involved in a managed treatment plan for pulmonary disease, hypertension (defined as systolic blood pressure consistently greater than 140 mm Hg and/or a diastolic blood pressure greater than 90 mm Hg), hepatorenal disease, musculoskeletal disorders, neuromuscular/neurological diseases, autoimmune diseases, cancer, peptic ulcers, or anemia;
8. I am medically prescribed by a physician to take or regularly take over the counter medications for any heart, pulmonary, thyroid, anti-hyperlipidemic, hypoglycemic, anti-hypertensive, endocrinologic (e.g. thyroid, insulin, etc.), neuromuscular/neurological, or androgenic medications due to possible further health hazards that could occur with diet alteration or exercise training;
9. I report any unusual adverse events associated with this study that in consultation with the study investigators or supervision physician recommends removal from the study;
10. I have taken ergogenic levels of nutritional supplements that may affect muscle mass or aerobic capacity (e.g., creatine, HMB) or anabolic/catabolic hormone levels (e.g., androstenedione, DHEA, etc.) within 6 months prior to the start of the study;
11. I have consumed any iron or mineral type dietary supplements (excluding multivitamins) 1 month prior to the study;
12. I have a history of food or drug allergy of any kind;
13. I have any other condition in which principal investigator thinks may jeopardize the study or the subject.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — A female participant who is aerobically trained (have a minimum of 42 ml/kg/min), between the age of 18 and 30 years.
Enrollment: 2 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-11-11 (Actual)

PRIMARY OUTCOMES:
Effect of IronAid IPS on Iron mcg/dL | 12 weeks (84 days)
  The primary purpose is to observe the effect of supplementation on fasting total iron levels prior to and after the supplementation period.
Effect of IronAid IPS on Ferritin ng/mL | 12 weeks (84 days)
  The primary purpose is to observe the effect of supplementation on ferritin levels prior to and after the supplementation period.
Effect of IronAid IPS on the Exercise Induced Feeling Inventory | 12 weeks (84 days)
  The primary purpose is to observe the effect of supplementation on feelings of fatigue prior to and after exercise testing in the laboratory at Week 0, 4, 12.
Effect of IronAid IPS on the Rate of Perceived Exertion Scale | 12 weeks (84 days)
  The primary purpose is to observe the effect of supplementation on feelings of fatigue after exercise testing in the laboratory at Week 0, 4, 12. The scale ranges from 6 to 20 with 6 labeled as "no exertion" and 20 labeled as "maximal exertion". All values are subjective and based on an individual's perception. For the purposes of this study, a value ranged as close to 20 as possible to ensure maximal effort is achieved.

SECONDARY OUTCOMES:
Effect of IronAid IPS on Glucose mg/dL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Urea Nitrogen (BUN) mg/Dl | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Creatinine mg/Dl | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on eGFR Non-Afr. American mL/min/1.73m2 | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on eGFR African American mL/min/1.73m2 | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on BUN/Creatinine Ratio calculated | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Sodium mmol/L | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Potassium mmol/L | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Chloride mmol/L | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Carbon Dioxide mmol/L | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Calcium mg/Dl | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Protein, Total g/Dl | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Albumin g/dL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Globulin g/Dl | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Albumin/Globulin Ratio calculated | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Bilirubin, Total mg/Dl | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Alkaline Phosphatase U/L | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Aspartate Aminotransferase U/L | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on Alanine Aminotransferase U/L | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of IronAid IPS on White Blood Cell Count thousand/uL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Red Blood Cell Count million/uL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Hemoglobin g/dL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Hematocrit % | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on MCV fL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on MCH pg | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on MCHC g/dL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on RDW % | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Platelet Count thousand/uL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on MPV fL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Absolute Neutrophils cells/uL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Absolute Lymphocytes cells/uL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Absolute Monocytes cells/uL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Absolute Eosinophils cells/uL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Absolute Basophils cells/uL | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Neutrophils % | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Lymphocytes % | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Monocytes % | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Eosinophils % | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on Basophils % | 12 weeks (84 days)
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of IronAid IPS on the Short form (36) Health Survey | Week 0, 4, 8, and 12
  The secondary purpose is to assess the effects of ingesting the supplement on the immune system by means of completing this survey at Week 0, 4, 8 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Lemuel W Taylor, PhD, Principal Investigator — UMHB Human Performance Lab
Locations (1):
- UMHB Human Performance Lab, Belton, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided